CLINICAL TRIAL: NCT04372693
Title: Unplanned Shifting the Traditional Classroom-Based to Online Distance Learning as a Result of (COVID-19) Social Distancing Measures: Nursing Students' Perception and Achievement
Brief Title: Unplanned Shifting to Online Distance Learning: Nursing Students' Perception and Achievement
Acronym: (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FON170133
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Distance Learning-Online Learning; Traditional Classroom-Based Learning; Coronavirus Disease Social Distancing Measures; Nursing Students' Perception and Achievement

STUDY DESIGN:
Intervention Model Description: Online Distance Learning with certain principals will be implemented for the study group and control group who learned by Traditional Classroom-Based will be selected retrospectively as baseline data, students' perception and achievement will be measured for both.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of students who are learning by Online Distance (Experimental): The following principals implemented while online learning will be processing;
  1. Address and consider the students' differences in online learning application as a new experience.
  2. Allow for Individual Locus of Control.
  3. Motivate the student:
  4. Avoid information overload,
  5. Create A real-life context,
  6. Encourage social interaction,
  7. Provide hands-on activities,
  8. Encourage student reflection.
  Interventions: Other: impliminting Online Distance Learning
- students who were learned by Traditional Classroom-Based (No Intervention)

INTERVENTIONS:
Other: impliminting Online Distance Learning — as a result of (COVID-19) social distancing measures, the Online Distance Learning will be implemented without prior planning for undergraduate nursing students
  Arms: group of students who are learning by Online Distance

SUMMARY:
Online Distance Learning (ODL) is an educational delivery system that helps students to join in an educational opportunity without physically existing in the same setting as the teacher. Online learning is known as the education that takes place over the Internet, often referred to as e-Learning, web-based training (WBT), distance learning, or asynchronous learning. When learners participate in an online learning course at different times, it is known as asynchronous learning. online learning involves the umbrella term for any learning that takes place across distance and not in a traditional classroom. WHO recommends Implement social distancing practices that may include; Staggering the beginning and end of the school day and Use of online/e-learning strategies? The coronavirus pandemic has changed how millions around the globe are educated. new shifts in education approaches could widen equality gaps. As of March 13, the Organization for Economic Co-operation estimated that over 421 million students are affected due to school closures announced or implemented in 39 countries. Most faculties in affected areas are finding stop-gap solutions to continue teaching, but the quality of learning is heavily dependent on the level and quality of digital access.

Therefore, the current study aimed to assess Nursing students' perception and achievement regarding unplanned shifting the Traditional Classroom-Based to Online Distance Learning as a result of (COVID-19) social distancing measures.

H1: Learning perception is lower for nursing students who learned by unplanned Online Distance Learning (μ1) than for those who learned by Traditional Classroom-Based learning (μ2), (H1: μ1 < μ2).

H1: Scholar achievement is greater for nursing students who learned by Traditional Classroom-Based learning (μ1) than for those who learned by unplanned Online Distance Learning (μ2), (H1: μ1 > μ2).

A quasi-experimental research design will be utilized in the current study with a comparative approach.

A purposive sample of adult male and female bachelor's students of nursing will be asked to participate in the current study.

Three tools will be adopted to collect data relevant to the current study.

1. A brief demographic self-administrated questionnaire
2. Students' Learning Perception Questionnaire (SLPQ),
3. Modified McVay's Readiness for Online Learning Questionnaire

DETAILED DESCRIPTION:
Online Distance Learning (ODL) is an educational delivery system that helps students to join in an educational opportunity without physically existing in the same setting as the teacher. Online learning is known as the education that takes place over the Internet, often referred to as e-Learning, web-based training (WBT), distance learning, or asynchronous learning. When learners participate in an online learning course at different times, it is known as asynchronous learning. Online learning involves the umbrella term for any learning that takes place across distance and not in a traditional classroom.

The reason for much of the growth in distance education programs in recent years is the development of the Internet and the improvement of technologies that support online learning environments. Despite the rapid growth in (OLD) use, there is a need to continuous assessment of its effectiveness. Numerous studies comparing traditional classroom-based instruction with technology-supported instruction have found no significant differences in critical educational variables such as learning outcomes and student satisfaction.

Students prefer certain methods of learning more than others. These traits, referred to as learning styles, form a student's unique learning preference, and aid teachers in the planning of small-group and individualized instruction. If optimal student learning is dependent on learning styles, and these styles vary between distance and equivalent on-campus students, then faculty should be aware of these differences and alter their preparation and instructional methods accordingly. Knowledge of student learning preferences can aid faculty in-class preparation, designing class delivery methods, choosing appropriate technologies, and developing sensitivity to differing student learning preferences within the distance education environment. Many communication skills required of the (ODL) instructor are similar to those needed for effective classroom teaching. On the other hand, the online instructor's role does require a paradigm shift regarding instructional time and space, virtual management techniques, and the ability to engage students through virtual communication.

The coronavirus pandemic has changed how millions around the globe are educated. WHO recommends implementing social distancing practices that may include; staggering the beginning and end of the school day and use of online/e-learning strategies . New shifts in education approaches could widen equality gaps. As of March 13, the Organization for Economic Co-operation estimated that over 421 million students are affected due to school closures announced or implemented in 39 countries. Besides, another 22 countries have announced partial "localized" closures. These risk-control decisions have led millions of students into temporary 'home-schooling' situations, these changes have certainly caused a degree of inconvenience, but they have also prompted new examples of educational innovation. To help slow the virus' spread, Academic 2.7 Million students in Egypt started to learning at home, in February 2020, via interactive apps, and other faculties got further simpler asynchronous online learning tools (such as reading material via Google Classroom, ZOOM, sending lessons and assignments via the official website, WhatsApp or email) augmented with synchronous face-to-face video instruction, to help preempt school closures.

Most faculties in affected areas are finding stop-gap solutions to continue teaching, but the quality of learning is heavily dependent on the level and quality of digital access. Moreover, the less affluent, digitally understanding, and low socioeconomic are factors affecting the student's achievement. For anyone who has taught face-to-face classes, making the transition to fully online may feel completely overwhelming. Course writers and instructors alike might find themselves asking questions such as, "How will I translate my classroom materials-activities or laboratory experiences-in a way that will benefit the online student? How will I generate discussion and engagement between students? Assessment of students' perception toward provided learning methods was growing in recent years because the best way of confirming quality in academic education is obtaining feedback from undergraduates . Many studies examined students' perception as a solo dimensional scale, such as self efﬁcacy, behavioral response, or effective response. While, in the current study the researcher prefers to utilize a comprehensive, widely used, valid, reliable, and multi-dimensional tool additionally avoid too-much items to prevent respondents fatigue.

Although the implementation of Online Distance Learning will be established as a result of (COVID-19) social distancing measures suddenly without any plan of action, one question remains a need for the answer; how prepared students are for successful Online Distance Learning? Whatever the answer may be, the new method of e-learning will be administrated for the student. The researcher believes that addressing the preparedness and rate the important competencies required by students for effective Distance Learning performance of the student is the first and important step. Although a number of the online learning readiness scales have been developed to assess the readiness of students to be online learners, very few of these scales provide an assessment concerning the knowledge, skills, and attitudes students might require as online learners. In many of the preparedness scales, there is the tendency to describe what students have to be (e.g., self-directed, self-aware) rather than what students need to do . In 2000, McVay developed a Readiness for Online Learning questionnaire that used attitudes and behaviors as predictors of online student learning readiness.

Therefore, the current study aimed to assess Nursing students' perception and achievement regarding unplanned shifting the Traditional Classroom-Based to Online Distance Learning as a result of (COVID-19) social distancing measures:

Theoretical framework Teachers must examine students' traditional perspectives and adopt a comprehensive perspective framework of learning environments that is appropriate for online teaching. Specific aspects of adult learning theory guided the development of the pedagogical model that was used to develop the online learning environment. Johnson, 1997 suggests a combination philosophy of learning theories rather than be confined to one preferred perspective such as; behavioral, Cognitive, and social learning theories. Quality online learning environments should be made up of elements of behavioral learning theory e.g. using positive reinforcement and repetition. Cognitive learning theory (for example, addressing Multiple senses, presenting new information in motivating ways, limiting the amount of information presented, and connecting new information to prior knowledge), and social learning theory (for example, encouraging group interaction, peer assessment, and personal feedback). These three theories were synthesized into integrated seven general principles that appear to be crucial for online learning environments. The current study adopting that the powerful online learning environments need to contain a combination of these principles: (1) address individual difference, (2) motivate the student, (3) avoid information overload, (4) create A real-life context, (5) encourage social interaction, (6) provide hands-on activities, and (7) encourage student reflection. These principles for online instruction will be attempted to apply all as a framework while facing the challenge of dramatical, situational, and unplanned application.

Research Hypothesis H1: Learning perception is lower for nursing students who learned by unplanned Online Distance Learning (μ1) than for those who learned by Traditional Classroom-Based learning (μ2), (H1: μ1 < μ2).

H1: Scholar achievement is grater for nursing students who learned by Traditional Classroom-Based learning (μ1) than for those who learned by unplanned Online Distance Learning (μ2), (H1: μ1 > μ2).

Subjects and Methods

Research Design:

A quasi-experimental research design will be utilized in the current study. The study group will be learned (prospectively) the selected courses by Online Distance method with following certain principles for effective online learning environments as a result of (COVID-19) social distancing measures in comparison to the control group of nursing students who (retrospectively) learned the same courses by the Traditional Classroom-Based learning. Both study and control groups will be assessed for students' perception and scholar achievement as a dependent effect. However, subjects of the current study will not randomly be assigned to either the experimental or the comparison group.

Participant:

A purposive sample of adult male and female bachelor's students of nursing who studying health assessment (clinical) and research in nursing courses will be asked to participate in the current study. The participant students will be divided into study and control groups. Students who studied in autumn Semester (Official started in September 2020) will be selected as a study group. While the control group will be selected as the students who studied the same courses in the autumn semester (started in 2019 September 21 to 2020 January 9). The estimated sample size is 180 participant, estimated by (G Power analysis) (independent t-tests - One tail, Effect size = 0.5, α = 0.05, Power (1-β) = 0.95, balanced allocation ratio 1:1). The students who studying the selected courses (expected to be 500 students) as well as have corresponding to the following inclusion criteria will included in the current study:

* None of the participants had previously taken the online-based course.
* The same educational background.
* Passed all pre- requisite courses.
* Full-time enrollment.

Instruments of Data Collection:

Three tools will be framed to collect data relevant to the current study.

1. A brief demographic self-administrated questionnaire was constructed to collect information on aspects such as the participant's gender, age group and enrollment level in addition to students' GPA, it will be collected from the student affairs of the college to measure the students' scholar achievement as a dependent variable.
2. Students' Learning Perception Questionnaire (SLPQ), will be utilized in the current study to measure students' perception as a dependent variable, (SLPQ) was adopted, inventory and metric instrument to assess the effectiveness of provided learning methods as perceived by the students, its reliable tool with Cronbach's Alpha 0.76 which reflect the degree of internal consistency among variables. It covers two inventories; students' perceptions of the teaching-learning environment (TLE) (22 items) and students' approaches to learning (SAL) (12 items). [12-13]. Six factors emerged from the 22 items measuring different aspects of the teaching-learning environment (TLE): (Teaching for understanding, Alignment, Staff enthusiasm, and support, Interest and relevance, Constructive feedback, and Support from other students). [14]. While, students' approaches to learning (SAL) measure three broad approaches to learning: deep approach to learning, surface approach to learning, and organized studying, each with four items. (SLPQ) Items will be scored on a five-point Likert scale ("Totally disagree (1)" to "Totally agree (5)") [12-14]. The scores of each students will be summed for interpretation, those who obtained less than (25%) will considered as having an low perception, while who obtained (26 - 75%) will considered as a moderate perception, and finally who get more than (75%) will considered as a high perception level.

   The instrument will be provided as its original language of English because the students learned and examined all courses in the English language. Arabic translation will be available to students if they faced difﬁculty in understanding any statement. Data will be collected from participants through an electronic questionnaire online using email (for control and experimental group).
3. Modified McVay's Readiness for Online Learning Questionnaire. Watkins et al. (2004) developed a 27 items adopted scale that used attitudes and behaviors of the participants as predictors of students' preparedness for online learning and e-learning environments, its reliable tool with Cronbach's Alpha 0.82. This self-administrated instrument identified six dimensions: Technology Access (3 items), Online Skills and Relationships (9 items), Motivation (3 items), Online Audio/Video (3 items), Internet Discussions (4 items) and Importance to your success (5 items). The instrument consisted of a 5-point Likert-type scale response format (1- Completely Disagree, 2-Strongly Disagree, 3- Not Sure, 4-Strongly Agree, 5-Completely Agree).

Ethical Consideration:

Participation in the study is voluntary; each participant has the right to withdraw from the study when he or she wants. Informed consent will be obtained from the participants. Confidentiality and anonymity of the subjects are assured through coding of all data. Collected data will be used for the research purpose only and will not be reused in another research. All information taken will be protected and will not affect students' annual appraisal by any means. The formulated database and the result of the current study will be incorporating into the plan of education in the college.

Procedure:

Once the official permission and ethical approval are granted to proceed to the proposed study, the implementation will be applied in two parts:

The first Part will be initiated by reviewing the selected students' data who are studying the selected courses in semester (autumn- 2019) and (autumn -2020). The contact information of the students who will correspond to the inclusion criteria will be obtained. Then, they will be invited by sent phone messages to participate in the current study. The student who willing to participate in this study will be divided into paired study and control groups. The students who will study in the (autumn- 2020) will be operated as a study group, also the students who are previously completed autumn 2019 semester will be manipulated as a control group. The excepted number of participants will be 500 students. The purpose, nature, and benefits of the study will be explained to the participants. A pilot study will be conducted on 10% = 18 students to estimate the needed time for data collection, and to test the feasibility, objectivity, and clarity of the study instruments. All queries of students regarding the meaning of the statements and how to ﬁll in the answers will be discussed via email and addressed before the actual study will start.

Second Part will be started by sending (instrument 1, 2) to the control group (students who were learned by Traditional Classroom-Based Learning) via electronic online survey system (Jot form) to fill out, the link of the created form was (https://www.jotform.com/help/408-understanding-your-account-usage-and-limits). These collected data will be considered as baseline data pertinent to the current study. About the study group (students who learned by online distance way) they will be asked first to fill out (instrument 1, 3) then, The following actions implemented while online learning will be processing;

(1) Address and consider the students' differences in online learning application as a new experience. Provide Content in Multiple Formats. use of various communication technologies. Lectures are audio streamed and synchronized with the applicable PowerPoint presentation. lectures are also transcribed and posted on the course Web site. Utilize links to outside Web sites that provide supplemental material on the current topic.

(2) Allow for Individual Locus of Control. Access the content through links or a graphical organizer. Access to organize the course material as students need. Students may even move through the course topics in random order.

* Encourage active and collaborative interaction. In light of the idea that the whole is greater than the sum of its parts, each course is designed with activities that are both individual- and group-based.

  (3) Motivate the student:
* Maintain students' attention by providing an environment that is engaging and participative. Make the students feel that the course material is relevant. Incorporate Games into the Online Environment. Use Multimedia When Appropriate.

  (4) Avoid information overload,
* Limit the Amount of Content and Number of Activities. Organize Instruction Around Learning Cycles. Provide a Graphic Organizer for the Course.

  (5) Create A real-life context,
* Create Virtual Learning Teams. Simulate Reality Using Appropriate Case Studies. Require Collaborative Projects (6) Encourage social interaction,
* Create a Personal Connection with Students. Peer Review and Feedback. Facilitate Interaction (7) Provide hands-on activities,
* Organize Online Courses Around Projects. Think-Pair-Share in a Virtual Environment. Use Small-Group Discussions During Synchronous Sessions.

  (8) Encourage student reflection.
* Provide Extensive and Timely Feedback and encourage online Diaries or Reflective Journals.

At the end of the current semester, the students of the study group will be asked to complete an electronic online survey system using (Jot form) (instrument 2). Also, the GPA of all participants in the study and control group will be collected from the student affairs. Finally, the researcher will compare the data of the study dependent variables to the collected baseline data (control group).

Data Analysis Upon completion of data collection, descriptive and inferential statistics will be utilized to test for differences among the study and control group subjects, using the SPSS program.

ELIGIBILITY:
Inclusion Criteria:

All students should have corresponded to the following inclusion criteria:

* None of the participants had previously taken the online-based course.
* The same educational background.
* Passed all pre-requisite courses.
* Full-time enrollment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Students' Learning Perception Questionnaire (SLPQ), | 1 month
  Electronic online Questionnaire will be utilized using (Jot form) the link of the created Questionnaire is https://www.jotform.com/help/408-understanding-your-account-usage-and-limits
  Students' Learning Perception Questionnaire (SLPQ), will be utilized in the current study to measure students' perception as a dependent variable, (SLPQ) was adopted, inventory and metric instrument to assess the effectiveness of provided learning methods as perceived by the students. It covers two inventories; students' perceptions of the teaching-learning environment (TLE) (22 items) and students' approaches to learning (SAL) (12 items) (SLPQ) Items will be scored on a five-point Likert scale rated from "totally disagree" (1)" to "Totally agree (5)") . students who obtained less than (25%) will be considered as having a low perception, while who obtained (26 - 75%) will be considered as a moderate perception, and finally who get more than (75%) will be considered as a high perception level.
students' scholar achievement. | 1 month
  students' GPA, it will be collected from the student affairs of the college to measure the students' scholar achievement as a dependent variable.

OTHER OUTCOMES:
Modified McVay's Readiness for Online Learning Questionnaire. | 1 month
  3- Modified McVay's Readiness for Online Learning Questionnaire.
  Electronic online Questionnaire will be utilized using (Jot form) the link of created Questionnaire is https://www.jotform.com/help/408-understanding-your-account-usage-and-limits
  Watkins et al. (2004) developed a 27 items adopted scale that used attitudes and behaviors of the participants as predictors of students' preparedness for online learning and e-learning environments, its reliable tool with Cronbach's Alpha 0.82. This self-administrated instrument identified six dimensions: Technology Access (3 items), Online Skills and Relationships (9 items), Motivation (3 items), Online Audio/Video (3 items), Internet Discussions (4 items) and Importance to your success (5 items). The instrument consisted of a 5-point Likert-type scale response format (1- Completely Disagree, 2-Strongly Disagree, 3- Not Sure, 4-Strongly Agree, 5-Completely Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Elhabashy, Lecturer, Principal Investigator — Faculty of Nursing-Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the study will be available to interested researchers by Publication in the indexed journal at the end of the study completion